CLINICAL TRIAL: NCT03642197
Title: Feasibility and Preliminary Efficacy of Support Figure Attendance at Bariatric Patients' Clinical Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Keeley Pratt, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0264
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Diet Habit; Behavior, Social; Physical Activity
Keywords: Bariatric Surgery; Obesity; Social Support; Health Behavior
MeSH Terms: conditions — Obesity, Morbid; Feeding Behavior; Social Behavior; Motor Activity; Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: A four-arm randomized controlled trial (RCT) using simple randomization will randomize female patients in romantic relationships into partner attended (PA) groups and treatment as usual (PA-TU) groups; patients (female or male) not in romantic relationships will be randomized into support figure attended (SFA) and SFA-TU groups.
  Patients in all arms will receive routine care. Support figures/partners of patients in the SFA and PA arms will be requested to attend the four pre-surgery classes with the patient and the three clinical visits; patients in the SFA-TU and PA-TU arms will attend individually.
  Assessments will be completed by patients and support figures/partners (all four arms) at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4). The study will follow all groups for roughly six months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Support Figure Attended (SFA) (Experimental): Using simple randomization patients (female or male) not in romantic relationships will be randomized into support figure attended (SFA) and SFA-TU groups. Patients in all arms will receive routine care, which includes four pre-surgery classes and routine clinical visits. Support figures in the SFA arm will be requested to attend the four pre-surgery classes with the patient and the three clinical visits. The intervention is support figure attendance. Assessments will be completed by patients and support figures at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4).
  Interventions: Behavioral: Attendance
- SFA - Treatment as Usual (SFA-TAU) (No Intervention): Using simple randomization patients (female or male) not in romantic relationships will be randomized into support figure attended (SFA) and SFA-TU groups. Patients in all arms will receive routine care, which includes four pre-surgery classes and routine clinical visits. Support figures in the SFA-TU arm will not be requested to attend the four pre-surgery classes with the patient and the three clinical visits- patients will attend alone. Assessments will be completed by patients and support figures at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4).
- Partner Attended (PA) (Experimental): Using simple randomization female patients in cohabiting romantic relationships for at least 6 months will be randomized into partner attended (PA) and PA-TU groups. Patients in all arms will receive routine care, which includes four pre-surgery classes and routine clinical visits. Partners in the PA arm will be requested to attend the four pre-surgery classes with the patient and the three clinical visits. The intervention is partner attendance. Assessments will be completed by patients and partners at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4).
  Interventions: Behavioral: Attendance
- PA - Treatment as Usual (PA-TAU) (No Intervention): Using simple randomization female patients in cohabiting romantic relationships for at least 6 months will be randomized into partner attended (PA) and PA-TU groups. Patients in all arms will receive routine care, which includes four pre-surgery classes and routine clinical visits. Partners in the PA-TU arm will not be requested to attend the four pre-surgery classes with the patient and the three clinical visits- patients will attend alone. Assessments will be completed by patients and partners at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4).

INTERVENTIONS:
Behavioral: Attendance — The SFA and PA arms will be instructed to attend pre-surgery classes and clinical visits with the patients.
  Arms: Partner Attended (PA); Support Figure Attended (SFA)

SUMMARY:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy for the inclusion of support figures and romantic partners throughout the bariatric surgery process, from pre-surgery to two months post-surgery. This will be done using a four-arm randomized controlled trial (RCT). Using simple randomization, female patients in romantic relationships will be randomized into partner attended (PA) groups and treatment as usual (PA-TU) groups; patients (female or male) not in romantic relationships will be randomized into support figure attended (SFA) and SFA-TU groups.

The goals of this study are to provide preliminary evidence for including support figures/partners in patients' routine BS healthcare visits, including the subsequent impact on post-surgery patient and support figure/partner behavior change and weight loss, relationship outcomes, and exploration of barriers to support figure/partner involvement.

Aim 1: To assess the feasibility and acceptability of support figure/partner involvement for BS patients. Feasibility will be assessed throughout the study by attendance at the four pre-surgery classes and the clinic visit assessment time points. Perceived fiscal and time involved in the study will be assessed. Acceptability will be assessed from patient and support figure/partner interviews regarding the barriers and benefits to attendance, and alternative mediums to engage support figures/partners.

Aim 2: To evaluate the effect of support figure/partner attendance (SFA, PA arms) on patient weight loss, behavior change, and relationship outcomes from T1-T4. Estimates of effect size and variance in patient weight loss and behavior change will be collected from T1-T4 for comparison of the SFA/PA and SFA-TU/PA-TU arms.

DETAILED DESCRIPTION:
The purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy for the inclusion of support figures and romantic partners throughout the bariatric surgery process, from pre-surgery to two months post-surgery. This will be done using a four-arm randomized controlled trial (RCT). Using simple randomization, female patients in romantic relationships will be randomized into partner attended (PA) groups and treatment as usual (PA-TU) groups; patients (female or male) not in romantic relationships will be randomized into support figure attended (SFA) and SFA-TU groups.

The goals of this study are to provide preliminary evidence for including support figures/partners in patients' routine BS healthcare visits, including the subsequent impact on post-surgery patient and support figure/partner behavior change and weight loss, relationship outcomes, and exploration of barriers to support figure/partner involvement.

Inclusion criteria for the PA arm requires patients be pre-surgery and registered for pre-surgery classes, identify as female, and in a romantic relationship with a cohabitating partner/spouse for at least 6 months. Inclusion criteria for the SFA arm requires patients be pre-surgery and registered for pre-surgery classes, and not be in a cohabitating romantic relationships. Known terminal illness diagnosis excludes patients and support figure/partner participation. The recruitment goal is 110 dyads in all four arms of the study (SFA, SFA-TU, PA, PA-TU).

Patients in all arms will receive routine care, which includes four pre-surgery classes and routine clinical visits. Support figures/partners of patients in the SFA and PA arms will be requested to attend the four pre-surgery classes with the patient and the three clinical visits; patients in the SFA-TU and PA-TU arms will attend individually. Assessments will be completed by patients and support figures/partners (all four arms) at the first pre-surgery class (T1) and routine clinical visits: the pre-surgery appointment (T2), two-weeks post-surgery appointment (T3), and at the two-months post-surgery appointment (T4).

Aim 1: To assess the feasibility and acceptability of support figure/partner involvement for BS patients. Feasibility will be assessed throughout the study by attendance at the four pre-surgery classes and the clinic visit assessment time points. Perceived fiscal and time involved in the study will be assessed. Acceptability will be assessed from patient and support figure/partner interviews regarding the barriers and benefits to attendance, and alternative mediums to engage support figures/partners.

Aim 2: To evaluate the effect of support figure/partner attendance (SFA, PA arms) on patient weight loss, behavior change, and relationship outcomes from T1-T4. Estimates of effect size and variance in patient weight loss and behavior change will be collected from T1-T4 for comparison of the SFA/PA and SFA-TU/PA-TU arms.

Hypothesis. Patients in the SFA and PA arms will experience increased weight loss, physical activity frequency, and higher compliance with post-surgery dietary recommendations compared to patients in the SFA-TU and PA-TU arms at T4.

Sub-aim 2.1. To evaluate the effect of attendance on support figure/partner weight status. Support figures and partners will complete measures of weight status at the same time points as the patient. Because it is largely unknown if support figures/partners could benefit from intervention with the patient, or if support figures/partners' weight status is similar to the patients, we will explore support figures/partners' weight status and if their weight status changes from T1 to T4.

Sub-aim 2.2. To determine the preliminary effect of attendance on relationship outcomes. Patients and support figures/partners will complete self-report measures of relationship quality (PA-only), attachment security (PA-only), family functioning, and perceived social support from T1-T4 to determine the effect of attendance on patient and support figure/partners' perspectives of relationship outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients in all arms must be ≥18 years-old, seeking bariatric surgery, speak and read/write English
* Partners and support figures must be ≥18 years old, speak and read/write English, and have no prior history of BS
* Partners in the PA and PA-TAU arms must be in a romantic relationship and cohabitate with the patient for at least 6 months

Exclusion Criteria:

* No known terminal health diagnosis (i.e., Cancer)
* In the PA and PA-TAU arms, no known domestic violence or abuse between partners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In the PA and PA-TAU arms, female patients will be recruited, partners can identify as male or female. In the SFA and SFA-TU arms patients identifying as male or female will be recruited, support figures can identify as male or female.
Enrollment: 63 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Percent Excess Weight Loss (%EWL, Patient) | 6 months, 4 time points
  [(T1 weight in lbs) - (Follow up (T2-T4) Weight)] / [(TI Weight) - (Ideal Weight)]

SECONDARY OUTCOMES:
Dietary Compliance (Patient) | 6 months, 4 time points
  Trained dieticians will conduct oral 24-hour recalls with patients and rate as (0) not compliant or (1) compliant. Ratings are based on the American Society of Metabolic Bariatric Surgery (ASMBS) surgery guidelines.
Physical Activity (Patient) | 6 months, 4 time points
  Scale Name: Bouchard's Physical Activity Record. Items 1-9 are totaled to assess physical activity intensity, ranging from 24-96, where higher scores indicate higher intensity of activity throughout the day.
Relationship Quality (Patient and Partner) | 6 months, 4 time points
  Scale Name: Abbreviated Dyadic Assessment Scale (ADAS). There are 7 items to assess relationship quality on a continuous scale from 0-35, where higher scores indicate higher relationship quality. Items are scored on a 0-5 scale for items 1-6, and 0-6 scale for item 7.
Perceived Social Support for Behavior Change (Patient and Partner/Support Figure) | 6 months, 4 time points
  Scale Name: Social Support for Eating Habits and Exercise. There are 23 items scored on a continuous scale ranging from 23-115 to assess perceived social support for behavior change, where higher scores indicate higher perceived support. Each item is scored on a scale ranging from 1-5. There are four subscales 1) encouragement of eating habits (items: 1-5); 2) discouragement of eating habits (6-10); and 3) family participation in exercise (items 11-16, 20-23); and 4) punishment for exercise (items: 17-19).

OTHER OUTCOMES:
Relationship Attachment (Patient and Partner) | 6 months, 4 time points
  Scale Name: Relationship Structures (ECR-RS) Questionnaire. There are 9 items averaged to assess relationship attachment on a scale of 1-7, where higher scores indicate higher avoidance or anxiety in the relationship. There are two subscales: 1) avoidance (items 1-6) and 2) anxiety (items 7-9). Items 1-4 are reversed.
Family Functioning (Patient and Partner/Support Figure) | 6 moths, 4 time points
  Scale Name: Family Assessment Device - General Functioning Subscale. There are 12 items assessed on a 1-4 scale, which are averaged to assess overall family functioning, where lower scores indicate healthier family functioning. There is an established clinical cut off score of 2.00, where scores at or above 2.00 indicate impaired family functioning. Odd numbered items are reverse coded.

CONTACTS AND LOCATIONS:
Overall Officials: Keeley J Pratt, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- Martha Morehouse Pavillion, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharpley, C. F., & Rogers, H. J. (1984). Preliminary validation of the Abbreviated Spanier Dyadic Adjustment Scale: Some psychometric data regarding a screening test of marital adjustment. Educational and Psychological Measurement, 44(4), 1045-1049.
- [Background] Fraley RC, Heffernan ME, Vicary AM, Brumbaugh CC. The Experiences in Close Relationships-Relationship Structures questionnaire: a method for assessing attachment orientations across relationships. Psychol Assess. 2011 Sep;23(3):615-25. doi: 10.1037/a0022898. PMID 21443364
- [Background] Epstein, N. B., Baldwin, L. M., & Bishop, D. S. (1983). The McMaster family assessment device. Journal of marital and family therapy, 9(2), 171-180.
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Bouchard C, Tremblay A, Leblanc C, Lortie G, Savard R, Theriault G. A method to assess energy expenditure in children and adults. Am J Clin Nutr. 1983 Mar;37(3):461-7. doi: 10.1093/ajcn/37.3.461. PMID 6829488